CLINICAL TRIAL: NCT06036017
Title: Determining the Effect of Care Package Implementation in Preventing Delirium in Patients Undergoing Coronary Artery Bypass Graft Surgery
Brief Title: Care Bundle's Impact on Delirium Prevention in CABG Patients
Acronym: CareBundle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: İslam Elagöz (Other)
Responsible Party: Sponsor-Investigator, İslam Elagöz, Principal Investigator, Kilis 7 Aralik University
Organization: Kilis 7 Aralik University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: kilis7Aralıkuniv
Record Dates: First submitted 2023-07-26; First posted 2023-09-13 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Delirium; Bypass Complication; Coronary Artery Bypass; Patient Care Bundles
Keywords: Coronary Artery Bypass Graft Surgery; Care bundle Application; Delirium Prevention; Postoperative Care; Cardiac Surgery; Intensive Care; Quality of Care; music
MeSH Terms: conditions — Delirium | interventions — Ear Protective Devices; Music Therapy

STUDY DESIGN:
Intervention Model Description: During T0 assessment, the TBF (Total Body Function), GCS (Glasgow Coma Scale), GKO (Glasgow-Koma Ölçeği), RCUO (Respiratory Care Unit Observation), RASS (Richmond Agitation-Sedation Scale), and CAM-ICU (Confusion Assessment Method for the Intensive Care Unit) forms will be completed for both groups of patients, and blood samples will be taken. During T1 assessment, the GCS, GKO, RCUO, RASS, and CAM-ICU forms will be completed for both groups of patients, and blood samples will be taken. Additionally, the duration of anesthesia, intubation, and sedation, as well as the amount of sedative drugs used, will be noted. The care package prepared for the study group will be applied by nurses working in the ward.At T2, the GCS, GKO, RCUO, RASS, and CAM-ICU forms will be completed for both groups of patients, and blood samples will be taken. The duration of stay in the intensive care unit will also be recorded.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control groups (No Intervention): T1: TBF, GCS, GKS, RCUOS, RASS, CAM-ICU forms will be filled out from the patients and blood samples will be taken.
  T2: GCS, GKS, RCUOS, RASS, CAM-ICU forms will be filled out from the patients and blood samples will be taken. Additionally, durations of anesthesia, intubation and sedation as well as the amount of medication used for sedation will be recorded. The care package prepared will be applied to this group by the nurses working at the ward.
  T3: GCS, GKS, RCUOS, RASS, CAM-ICU forms will be filled out from the patients and blood samples will be taken. Their length of stay in the intensive care unit will be noted.
- Study groups (Experimental): T1: TBF, GCS, GKS, RCUOS, RASS, CAM-ICU forms will be filled out from the patients and blood samples will be taken.
  T2: GCS, GKS, RCUOS, RASS, CAM-ICU forms will be filled out from the patients and blood samples will be taken. Additionally, durations of anesthesia, intubation and sedation as well as the amount of medication used for sedation will be recorded.
  T3: GCS, GKS, RCUOS, RASS, CAM-ICU forms will be filled out from the patients and blood samples will be taken. Their length of stay in the intensive care unit will be noted.
  Interventions: Other: Earplugs; Other: Music Therapy; Other: Presence of Family After Extubation:

INTERVENTIONS:
Other: Earplugs — There are numerous studies that suggest using earplugs can regulate a patient's sleep and may reduce the risk of delirium (Locihova 2017) (Van Rompaey 2012). However, there is no hard and fast rule concerning the duration, timing, and preference of earplug use. The duration of earplug use may vary and will be determined based on the needs of the patient, and it will be ensured that they are used throughout the night (Rompaey 2012).
  Arms: Study groups
Other: Music Therapy — Music therapy will be applied to help the patient relax and fall asleep. Moreover, the choice of music genre will be suitable for the patient's preferences, and it will be ensured that it is played at a low volume. Specific guidelines will be applied regarding the frequency and duration of music therapy, it will be performed twice a day after surgery at a low volume and via headphones, each session lasting 30 minutes (Sibenda A et al. 2019).
  Arms: Study groups
Other: Presence of Family After Extubation: — According to the guidelines titled 'Family presence and visit in Adult ICU' published by the American Association of Critical Care Nurses (AACN) in 2012; it is recommended that a family member or friend chosen by the patient be present to provide 24-hour uninterrupted emotional and social support for patients in intensive care. Allowing the patient's family to visit helps maintain the patient's social connections and contributes to the psychological well-being of the patient with family support. In addition to routine visits, patients' families can spend longer periods with the patient during their intensive care process and information about the patient is conveyed to close family members. Research shows that family presence in the intensive care unit reduces the incidence of delirium (Eghbali-Babadi, 2017) (Rosa 2017).
  Arms: Study groups

SUMMARY:
This research investigates the effectiveness of a care package used in the care of patients undergoing coronary artery bypass graft (CABG) surgery in preventing postoperative delirium. CABG surgery is a common procedure used to increase blood flow to the heart and is typically applied in patients with severe cardiac diseases. However, this procedure can increase the risk of postoperative delirium, especially among elderly and critically ill patients.

In this study, the goal is to reduce this risk by implementing a care package. The care package includes optimal pain management, sleep regulation, mobilization, ensuring patient orientation, and appropriate medication management.

The results of the research will be used to determine whether the use of this care package is effective in reducing the risk of delirium after CABG surgery. This could potentially improve patient outcomes and allow for more efficient use of hospital resources.

DETAILED DESCRIPTION:
Open-heart surgery is an effective treatment method used in the treatment of heart diseases today. However, after this operation, patients are at risk of postoperative delirium, which negatively affects the patient's recovery process. Open-heart surgery is a commonly performed surgical procedure; despite technological advancements and improvements in hospital care, delirium after open-heart surgery remains a common complicationDelirium, a condition causing acute dysfunction in the brain, leads to changes in patients' mental states and impairments in cognitive functions. Delirium after open-heart surgery is a common complication and can increase the patient's morbidity and mortality. Delirium extends the hospital stay and increases patient care costs. Therefore, it is important to implement a special care package to reduce the risk of delirium. The frequency of delirium in patients undergoing open-heart surgery varies between 20% and 50%. The post-open-heart surgery delirium prevention care package is a series of practices designed to reduce the patient's delirium risk. These practices may include; maintaining a regular sleep pattern, noise control, balancing hormone levels, family proximity, and music therapy.

Antipsychotic drugs, a pharmacological agent, are commonly used in the treatment of delirium. These drugs help to alleviate the symptoms of delirium and make the patient more calm. However, antipsychotic drugs are effective in symptom management and their side effects worsen the patient's condition and the effectiveness of antipsychotic drugs on delirium is doubtful. It is extremely important to avoid routine application of antipsychotic drugs. Instead, non-pharmacological methods are preferred, such as providing a suitable environment, regulating noise and light levels, maintaining sleep patterns, increasing physical activity, preventing unnecessary drug use, and regulating fluid and electrolyte balance. These methods can reduce the risk of delirium and help the patient undergo a faster and more successful recovery process.

There is a significant place in the literature for non-pharmacological methods for the prevention of delirium. These methods include ensuring the suitability of the environment the patient is in, regulating sleep schedules, keeping noise and light levels under control, psychological support and rehabilitation, pain and symptom management, prevention of sensory disorders, reducing invasive procedures, increasing physical activity, encouraging sleep, preventing unnecessary drug use, family-centered care, regulating fluid and electrolyte balance, and arranging nutritional order. The implementation of these methods can help avoid delirium risk factors and contribute to a faster recovery process for the patient.

Delirium is a very distressing condition for family members, especially those who observe delirium attacks. This situation can also have lasting effects on patients who remember delirium attacks in the hospital. It can also cause difficulties for the healthcare personnel caring for these patients. Therefore, it is extremely important to take the best possible precautions against delirium attacks or to treat the disease.

Family-centered care is an important factor in reducing the risk of delirium in patients during the postoperative period. Family members can be by the patients' side, provide moral support, and help patients feel more peaceful and comfortable in the postoperative period. Family members' support can reduce the patient's delirium risk, as it helps the patient maintain a familiar environment. A support network can also be critical in observing symptoms of delirium and ensuring appropriate treatment is sought.

Involvement of family members in patient care can be beneficial in many ways. For example, they can help orient the patient to time, place, and situation, provide emotional support, and communicate the patient's needs and preferences to the healthcare team. They can also encourage the patient to engage in physical activity, eat, and drink, which can help maintain their overall health and well-being.

Music therapy, one of the non-pharmacological methods, is also known to be effective in preventing delirium after open-heart surgery. Music therapy can help to reduce anxiety and promote relaxation, both of which can aid in delirium prevention.

In addition to these, maintaining a regular sleep pattern, controlling noise levels, and balancing hormone levels can be very effective in reducing the risk of delirium. Disruptions in sleep can lead to a higher risk of delirium, so ensuring the patient has a quiet and calm environment for rest can be crucial.

In conclusion, prevention of delirium after open-heart surgery is vital for the successful recovery of patients. A multi-faceted approach that includes non-pharmacological interventions such as environmental modifications, family-centered care, music therapy, and maintaining a regular sleep pattern, in addition to pharmacological treatments when necessary, is likely to be most effective. Further research is needed to identify the most beneficial and feasible interventions for preventing delirium after open-heart surgery.

ELIGIBILITY:
Inclusion Criteria:

Participants and Sample Criteria Inclusion criteria for the study:

* Over 18 years of age,
* Considered as a low-risk group according to American Society of Anesthesiologists (ASA)
* I-II and EUROSCORE scores
* Undergoing open-heart surgery for the first time
* Having an operation with on-pump and median sternotomy technique,
* Mild and moderate hypothermia applied,
* One to three coronary artery bypass grafts performed,
* Left internal mammary artery and saphenous vein graft applied,
* Surgery initiated between 08:00-12:00 hours,
* Having no psychiatric diagnosis and therefore no drug therapy,
* Not using corticosteroid derivative drugs,
* No complications observed that may affect the surgery and ICU process,
* Having a family member who can support the patient in the postoperative wake-up process,
* Patients who voluntarily agree to participate in the research will be included.

Exclusion Criteria:

* Extended surgery due to complications,
* Completion of the intraoperative process falls into the evening hours (after 16:00),
* Consciousness level after extubation prevents participation in the study (Glasgow Coma Score <15),
* Corticosteroid derivative drugs applied at any stage of the perioperative process, Surgery is canceled,
* No family member is available to stay in the intensive care unit,
* Wishing to withdraw from the research at any stage after voluntarily agreeing to participate in the study,
* At any stage of the research, patients who do not wish to use earplugs or listen to music and wish to withdraw from the research, their data will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
1.Introductory Information Form | up to 12 months
  This form comprises 21 closed-ended questions inquiring about age, gender, height, weight, educational level, employment status, the reason for applying to the cardiology surgery clinic, the year of heart disease diagnosis, presence of accompanying chronic diseases, previous surgery status, and dependency status.
2.Glasgow Coma Scale (GCS) | up to 12 months
  The Glasgow Coma Scale (GCS) is the most frequently used scale to evaluate the level of consciousness and was developed in 1974. It is used in emergency departments and intensive care units. The GCS consists of three sections that assess eye response, motor response, and verbal response. The total score ranges between 3 and 15, with scores between 13-15 indicating alertness, 8-12 suggesting a pre-coma state, and scores below 8 indicating a coma. However, it has some limitations, such as inadequacies in evaluating the verbal score of unconscious patients and the inability to assess parameters providing information about the depth of the coma. Nevertheless, it is widely used.
Visual Analogue Scale (VAS) | up to 12 months
  The Visual Analog Scale (VAS) is a method used to determine the intensity of pain, allowing patients to express their pain levels numerically. The full title of the scale is "Visual Analog Scale". This scale ranges from 0 to 10, with 0 indicating no pain and 10 representing the most intense pain. Higher scores indicate more severe pain. This method simplifies the definition of pain intensity and facilitates scoring and recording for health professionals. The scale provides guidance in evaluating ceiling and floor effects and is considered a reliable method for postoperative pain assessment. This method is used in numerous national and international studies and is included in current guidelines. Therefore, the choice to use this scale in pain intensity assessment is based on its reliability and widespread use.
Richard-Campbell Sleep Scale (RCSS): | up to 12 months
  This scale was developed by Richards and consists of six different criteria examining the depth of nighttime sleep, time to fall asleep, frequency of awakening, duration of wakefulness, quality of sleep, and the level of ambient noise. Each criterion is assessed on a scale ranging from 0 to 100. The scale's scoring system represents very poor sleep with scores between "0-25" and very good sleep with scores between "76-100." However, the sixth item measuring ambient noise level is excluded from the overall scoring, and the total score is calculated based on the five criteria. The higher the scale score, the better the patient's sleep quality. The validity and reliability of this scale is determining a Cronbach α value of 0.91. This value indicates high internal consistency of the scale.
Richmond Agitation-Sedation Scale (RASS) | up to 12 months
  RASS, developed by Cook and Palma in 1989 and introduced by Sessler in 2002, is designed specifically to determine the levels of sedation (calming) and agitation (restlessness) in ICU patients. RASS uses a 10-point scale to indicate levels of anxiety and agitation (+1 to +4 [combative]), a calm and awake state (0), and a state where the patient cannot be awakened (-5). The scale is designed with a central anchor at level 0, positive numerical grades for agitation, and negative numerical grades for sedation.
Confusion Assessment Method for the Intensive Care Unit (CAM-ICU): | up to 12 months
  Developed by Ely and colleagues in 2001, this scale underwent validity and reliability tests for internal and coronary ICU patients, demonstrating a sensitivity of 93-100% and specificity of 98-100%. A Turkish validity and reliability study conducted by Akıncı and colleagues in 2005 showed that the use of this scale in nursing observations could assist in the early diagnosis of delirium in the ICU and in taking preventive measures before treatment. However, factors such as patient age, level of consciousness, and disease prognosis can create disadvantages during diagnostic evaluation. In CAM-ICU, consciousness assessment is done in two steps. Step 1 evaluates the sedation state with the Richmond Agitation-Sedation Scale (RASS), while Step 2 uses CAM-ICU to determine symptoms of delirium.
Maintenance Package Checklist: | up to 12 months
  The maintenance package implementation checklist will be created by an interdisciplinary team, gathering evidence-based high-level applications from the literature. This list will carefully include a total of 4 items chosen to reduce the risk of delirium in patients during the postoperative period and to ensure they receive high-quality care. This list, crafted by expert teams, will be used by healthcare professionals to enhance patient outcomes.
Delirium Preventive Care Package Compliance Schedule | up to 12 months
  The compliance monitoring schedule will indicate on which days individuals will observe the adherence of healthcare professionals to the care package. For this purpose, a compliance tracking schedule will be prepared, and health professionals will follow this on specified days. The monitoring schedule will be arranged according to the working hours of health professionals ensuring they can access it at appropriate times. Thus, healthcare professionals, who are informed about the necessity of implementing the care package, will follow the compliance schedule, ensuring the successful progression of patient treatment. The compliance schedule will also help both health professionals and patient relatives feel confident that the care package is being regularly monitored.

CONTACTS AND LOCATIONS:
Overall Officials: İslam Elagoz, Ress. ass., Study Chair — kilis 7 Aralik Univ.
Locations (1):
- Islam, Kilis, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) collected in this study will be stored and processed in accordance with privacy and data protection laws. It is not planned to share these data with third parties. This policy is intended to protect the privacy and security of participants' personal information.